CLINICAL TRIAL: NCT05130840
Title: Feasibility of Multi-modality Central Nervous System Evaluation in HER2+ Breast Cancer Patients
Brief Title: Monitoring for Cancer Spread to the Central Nervous System (CNS) in People With Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-440
Record Dates: First submitted 2021-11-22; First posted 2021-11-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Central Nervous System; HER2+ Breast; 21-140
MeSH Terms: conditions — Breast Neoplasms | interventions — Spinal Puncture

STUDY DESIGN:
Intervention Model Description: This represents a two-cohort feasibility study to establish the feasibility of a multi-modality central nervous system (CNS) disease detection platform in patients with HER2+ breast cancer with no known CNS metastatic disease. Patients will enroll into one of 2 cohorts. Cohort A will be open to patients with Stage IV HER2+ breast cancer and Cohort B will include patients with Stage II-III HER2+ breast cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage IV HER2+ breast cancer (Experimental): Once enrolled on study, patients will undergo screening MRI Brain (unless already done as standard of care within 2 months on enrollment to evaluate for CNS disease) as well as lumbar puncture to evaluate for CNS disease. Once on study, patients will undergo LP and MRI Brain at 2 timepoints 6 months apart (+/- 8 weeks). LP will be performed to analyze cerebrospinal fluid for: cytology, circulating tumor cells and cell-free DNA. 6-month intervals for investigations have been based on feedback from patient advocates as well as clinical determination.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Lumbar puncture
- Stage II-III HER2+ breast cancer (Experimental): Once enrolled on study, patients will undergo screening MRI Brain (unless already done as standard of care within 2 months on enrollment to evaluate for CNS disease) as well as lumbar puncture to evaluate for CNS disease. Once on study, patients will undergo LP and MRI Brain at 2 timepoints 6 months apart (+/- 8 weeks). LP will be performed to analyze cerebrospinal fluid for: cytology, circulating tumor cells and cell-free DNA. 6-month intervals for investigations have been based on feedback from patient advocates as well as clinical determination.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Lumbar puncture

INTERVENTIONS:
Diagnostic Test: MRI — MRI Brain (unless already done as standard of care within 2 months on enrollment to evaluate for CNS disease) MRI Brain at 2 timepoints 6 months apart (+/- 8 weeks).
Diagnostic Test: Lumbar puncture — LP at 2 timepoints 6 months apart (+/- 8 weeks). LP will be performed to analyze cerebrospinal fluid for: cytology, circulating tumor cells and cell-free DNA.

SUMMARY:
The researchers doing this study think that performing scans of the brain and testing cerebrospinal fluid (CSF) in people with HER2-positive breast cancer may be an effective way of identifying the early onset of CNS metastases (such as brain cancer). If the researchers can identify the early onset of CNS metastases, they can immediately treat that cancer and possibly prevent it from worsening. Currently, people with breast cancer don't usually have scans of the brain or CSF testing unless they are experiencing symptoms of CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IV metastatic HER2+ breast cancer without CNS disease s/p 1 or more lines of HER2 directed therapy (Cohort A Only)
* Patients with Stage II-III HER2+ breast cancer without CNS disease (Cohort B Only)
* Male and Female participants Age ≥18 years
* HER2+ as defined by ASCO/CAP guidelines*
* Ability to undergo bedside Lumbar puncture to obtain cerebrospinal fluid; if beside LP is not successful due to patient discomfort or inability to obtain spinal fluid then patients will be offered LP through interventional radiology and patients will continue to be monitored on study
* Patients with breast implants and/or tissue expanders are eligible if they are able to safely undergo an MRI
* Able to provide written informed consent *ASCO/CAP guidelines: HER2+ defined as IHC 3+ positive and/or by ISH average copy number ≥ 6 signals/cell

Exclusion Criteria:

* Patients who are unable to undergo MRI with gadolinium
* Patients with CNS Metastases on Screening MRI
* Patients with Positive Cytology on Screening Bedside lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of eligible patients completing initial MRI | 2 years
  will require 8 out of 10 eligible patients to successfully complete the initial MRI
Percentage of eligible patients completing cerebrospinal fluid (CSF) evaluation | 2 years
  will require 8 out of 10 eligible patients to successfully complete the CSF evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wilcox, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm